CLINICAL TRIAL: NCT03527342
Title: Sahlgrenska University Hospital Cardiomyopathy Project: Mapping and Diagnosis of Cardiomyopathies to Enable Early and Specific Treatment
Brief Title: Sahlgrenska Cardiomyopathy Project
Status: Enrolling by invitation | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SUCARD
Record Dates: First submitted 2018-04-23; First posted 2018-05-17 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Dilated Cardiomyopathies; Hypertrophic Cardiomyopathy; Restrictive Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy; Myocarditis; Sarcoidosis With Myocarditis; Giant Cell Myocarditis; Amyloidosis; Heart (Manifestation)
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Restrictive; Arrhythmogenic Right Ventricular Dysplasia; Myocarditis; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Dilated Cardiomyopathy
- Myocarditis
- Sarcoidosis Heart
- Giant Cell Myocarditis
- Amyloidosis Heart
- Hypertrophic Cardiomyopathies
- Left Ventricular Myocardial Noncompaction Cardiomyopathy
- Arrhythmogenic Right Ventricular Cardiomyopathies

SUMMARY:
This is a joint project by Sahlgrenska University Hospital: Sahlgrenska, Östra and Mölndal.

Our objective is to diagnose and map patients with well phenotyped cardiomyopathies (CMP) including in depth clinical and molecular phenotyping to enable earlier and specific treatment. The project will serve as:

1. resource for diagnostic and therapeutic trials
2. common biomaterial bank
3. resource for detailed molecular analyses on patients' biomaterials and patient specific symptoms and examination results

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary cardiomyopathies including hereditary and inflammatory dilated cardiomyopathy, hypertrophic cardiomyopathy, restrictive cardiomyopathy, left ventricular non-compaction cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, myocarditis, giant cell myocarditis, sarcoidosis and amyloidosis engaging the heart

Exclusion Criteria:

* Patient with other preexisting cardiac diseases such as significant valvular, ischemic or pericardial disease before they receive a cardiomyopathy diagnose
* patients < 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are all patients referred to Sahlgrenska University Hospital, Gothenburg, Sweden with a cardiomyopathy diagnose.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression | 2018-2028

OTHER OUTCOMES:
Progression in biomarker NT-proBNP | 2018-2028
Changes over time in presence of autoantibodies | 2018-2028
Disease activity evaluated by positron-emissions-tomography computed tomography (PET-CT) | 2018-2028
Disease activity evaluated by magnetic resonance imaging (MRI) | 2018-2028

CONTACTS AND LOCATIONS:
Locations (1):
- Göteborg University, Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No